CLINICAL TRIAL: NCT00931879
Title: The Role of Lovaza® on Microvascular Function and Lipoprotein Profile in Type 2 Diabetes
Brief Title: Lovaza® and Microvascular Function in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Aaron I. Vinik, MD, PhD, Principal Investigator, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LVZ111903
Record Dates: First submitted 2009-06-17; First posted 2009-07-02 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Hypertriglyceridemia; Diabetic Neuropathy
MeSH Terms: conditions — Hypertriglyceridemia; Diabetic Neuropathies | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects are males or non-pregnant, non-lactating females age 18-80 years. All subjects must have been diagnosed with type 2 diabetes mellitus a minimum of two years according to the current ADA criteria and triglyceride levels above 149 mg/dL. Subjects in this arm will be taking placebo for 6 months.
  Interventions: Drug: Placebo
- omega-3-ethyl esters 4g (Active Comparator): Subjects are males or non-pregnant, non-lactating females age 18-80 years. All subjects must have been diagnosed with type 2 diabetes mellitus a minimum of two years according to the current ADA criteria and triglyceride levels above 149 mg/dL. Subjects in this arm will be taking 4 g of Lovaza per day for 6 months.
  Interventions: Drug: omega-3-ethyl esters

INTERVENTIONS:
Drug: omega-3-ethyl esters — Lovaza (TM) (omega-3-ethyl esters) 1 gram Capsules are indicated as an adjunct to diet to reduce very high (>500 mg/dL) triglyceride (TG) levels in adult patients.
  Other Names: Lovaza
  Arms: omega-3-ethyl esters 4g
Drug: Placebo — Subjects are males or non-pregnant, non-lactating females age 18-80 years. All subjects must have been diagnosed with type 2 diabetes mellitus a minimum of two years according to the current ADA criteria and triglyceride levels above 149 mg/dL. Subjects in this arm will be taking placebo for 6 months.
  Arms: Placebo

SUMMARY:
The objective of this study is to determine the efficacy of 6 months of 4 g/day oral Lovaza® on endothelial-dependent and heat-induced vasodilation in type 2 diabetics with neuropathy and elevated triglyceride levels. Omega-3 fatty acids appear to exert beneficial effects on vascular function that are independent of the changes in serum triglycerides. The efficacy will be compared with a placebo given at the same duration. Efficacy of the drug will be evaluated after 3 and 6 months of treatment. This timeline should be adequate for evaluation of the primary neurophysiological endpoints. Previously, the investigators have demonstrated that it is feasible to pharmacologically alter nerve fiber density in as little as 18 weeks and that this correlates with subjective and objective measures of neurovascular function. The investigators are predicting an enhancement of post-ischemic hyperemia of the foot dorsum, where the dilative mechanism is primarily endothelium-dependent and a similar improvement in heat-induced hyperemia.

DETAILED DESCRIPTION:
This pilot study is a within-subject repeated measures design. This study will compare the neurophysiological and vascular responses to placebo and treatment with Lovaza® (omega-3-acid ethyl esters, Reliant Pharmaceuticals, Inc.) in subjects with type 2 diabetes, neuropathy, and dyslipidemia.

Lovaza's potential mechanism of action is the inhibition of acyl Coenzyme A:1, 2-diacylglycerol acyltransferase and increased peroxisomal β-oxidation in the liver.

Subjects will be recruited and a baseline of physiological, neurological and hematological profile established for each patient. Forty-four subjects (20 in the active arm, 20 in the placebo arm, and 2 replacements for each arm) will receive 4 g/day Lovaza® tablets or placebo for a period of 6 months. All subjects will receive a physical and neurological exam as well as neurovascular function testing. This includes nerve conduction studies, quantitative sensory testing, quantitative autonomic testing, and skin blood flow testing, which includes, ischemia reperfusion. Lab tests include an insulin resistance profile, hepatic and renal function profiles, lipid profile, C-reactive protein, thyroid stimulating hormone, and fatty acids. Other tests include inflammatory markers such as adiponectin and tumor necrosis factor-α. The study is powered to detect differences in microvascular function after 6 months of Lovaza® and differences in ethnic responses.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects may be males or non-pregnant, non-lactating females age 18-80 years.
2. Subjects must have been diagnosed with type 2 diabetes mellitus according to the current ADA criteria.
3. Triglyceride levels above 149 mg/dL
4. Minimum of 2 years after diagnosis of type 2 diabetes
5. Prior to participation in this study, each subject must sign an informed consent document.

Exclusion Criteria:

1. Presence of type 1 diabetes mellitus (defined as C-peptide < 1 ng/ml or diabetes onset at < 35 years of age in a non-obese patient).
2. Presence of diabetic retinopathy that is more severe than "background" level.
3. Presence of diabetic nephropathy, defined by urine dipstick results greater than 300 mg/100 mL for protein (proteinuria).
4. Presence of clinically significant neuropathy that is clearly of non-diabetic origin, e.g. alcoholic or autoimmune.
5. Bilateral amputation of lower extremities or foot ulcers involving the great toes. Presence of neuroarthropathy (Charcot deformity) is allowable.
6. History of major macrovascular events such as myocardial infarction or stroke.
7. Participation in another clinical trial concurrently or within 30 days prior to entry into this study.
8. The use of ACE-inhibiting agents or angiotensin receptor blockade therapy (ARB) is allowed but must have been stable for at least 30 days prior to study entry and may not change during the course of the study. This is prudent due to their potential effects on blood flow.
9. Patients with moderate or severe hepatic insufficiency or abnormalities of liver function defined as any liver enzymes (aspartate aminotransferase,alanine transaminase, alkaline phosphatase) greater than 3 times the upper limit of normal.
10. Presence of pedal edema.
11. Presence or history of heart failure New York Heart Association Class II or greater.
12. Other serious medical conditions that in the opinion of the investigator, would compromise the subject's participation in the study.
13. Concomitant use of medications known to exacerbate triglyceride levels, such as estrogens.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron I Vinik, MD, PhD, Principal Investigator — Eastern Virginia Medical School; Henri K Parson, PhD, Study Director — Eastern Virgina Medical School
Locations (1):
- Strelitz Diabetes Center, Norfolk, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lovaza: Subjects are males or non-pregnant, non-lactating females age 18-80 years. All subjects must have been diagnosed with type 2 diabetes mellitus a minimum of two years according to the current ADA criteria and triglyceride levels above 149 mg/dL. Subjects in this arm will be taking 4 g of Lovaza per day for 6 months.
  omega-3-acie ethyl esters: Lovaza (TM) (omega-3-ethyl esters) 1 gram Capsules are indicated as an adjunct to diet to reduce very high (>500 mg/dL) triglyceride (TG) levels in adult patients.
Period: Overall Study
Arm/Group | Placebo | Lovaza
Started | 22 | 22
Completed | 19 | 19
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Population: The study was powered at 0.80 for a two-tail analysis with a sensitivity of a 30% delta in blood flow in 40 subjects. The standard deviation of the measurements was calculated at 45% of the treatment group mean. This assessment of variance could accommodate for 9% attrition or data loss in the study. 44 patients will be recruited in total.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lovaza | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.58 (2.06) | 58.21 (1.70) | 59.39 (1.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 17 | 17 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Weight (lbs) [Mean (Standard Deviation); unit: lbs] | 217.03 (9.62) | 215.16 (10.38) | 215.71 (7.25)
BMI kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 34.04 (1.17) | 34.37 (1.83) | 34.10 (1.11)
Qualifying triglyceride level (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 215.05 (12.51) | 261.17 (50.73) | 237.48 (24.42)
Total cholesterol (mg/dL) [Mean (Standard Deviation); unit: (mg/dL)] | 152.26 (6.56) | 189.42 (9.63) | 170.84 (6.51)
HDL cholesterol (mg/dL) [Mean (Standard Deviation); unit: (mg/dL)] | 39.84 (2.27) | 43.32 (2.81) | 41.58 (1.80)
LDL cholesterol (mg/dL) [Mean (Standard Deviation); unit: (mg/dL)] | 75.84 (5.80) | 101.44 (7.21) | 88.30 (5.01)
HbA1c (%) [Mean (Standard Deviation); unit: %] | 7.82 (0.35) | 7.66 (0.23) | 7.73 (0.21)
Fasting glucose (mg/dL) [Mean (Standard Deviation); unit: (mg/dL)] | 155.89 (9.18) | 157.21 (12.09) | 156.55 (7.49)
serum glutamate oxaloacetate transaminase(AST) (u/L) [Mean (Standard Deviation); unit: (u/L)] | 22.16 (1.50) | 24.11 (2.28) | 24.00 (8.44)
serum glutamate pyruvate transaminase (ALT) (u/L) [Mean (Standard Deviation); unit: (u/L)] | 28.79 (2.63) | 31.05 (3.84) | 30.71 (2.20)
Alkaline phosphatase (u/L) [Mean (Standard Deviation); unit: (u/L)] | 77.89 (6.55) | 70.11 (4.40) | 74.63 (4.62)
C-peptide (ng/mL) [Mean (Standard Deviation); unit: (ng/mL)] | 4.66 (0.40) | 4.56 (0.45) | 4.61 (0.30)
Insulin (uIU/mL) [Mean (Standard Deviation); unit: (uIU/mL)] | 39.54 (12.63) | 26.23 (5.88) | 32.88 (6.96)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Measures Are Nerve Conduction Studies, Specifically Changes in Conduction Amplitude.
Description: 19 participants in each arm( placebo or omega-3-ethyl esters 4g) were analyzed . Conduction velocities and amplitude of the following nerves were compared between each arm: Tibial Nerve Ankle Amplitude, Tibial Nerve Popliteal Amplitude, Median Nerve Wrist Amplitude, Median Nerve Elbow Amplitude, Peroneal Motor Nerve Ankle Amplitude, Peroneal Motor Nerve Below Fibular Amplitude, Peroneal Motor Nerve Above Fibular Amplitude, Sensory Median Nerve Wrist Amplitude, Sensory Ulnar, Sensory Sural Ankle Ampltiude Wrist Ampltiude
Time Frame: One year
Measure: Mean (Standard Error); unit: uV
Arm/Group | Placebo | Omega-3-ethyl Esters 4g
Number analyzed (Participants) | 19 | 19
uV
  Tibial Nerve Ankle Amplitude | 7.28 (0.94) | 7.14 (1.13)
  Tibial Nerve Popliteal Amplitude | 4.08 (0.58) | 3.80 (0.73)
  Median Nerve Wrist Amplitude | 6.89 (0.60) | 7.24 (0.55)
  Median Nerve Elbow Amplitude | 5.21 (0.56) | 6.06 (0.58)
  Peroneal Motor Nerve Ankle Amplitude | 2.97 (0.47) | 2.55 (0.36)
  Peroneal Motor Nerve Below Fibular Amplitude | 2.70 (0.46) | 2.17 (0.32)
  Peroneal Motor Nerve Above Fibular Amplitude | 2.79 (0.46) | 2.11 (0.31)
  Sensory Median Nerve Wrist Amplitude | 22.96 (3.04) | 26.56 (5.09)
  Sensory Ulnar Wrist Ampltiude | 26.93 (3.39) | 21.65 (5.13)
  Sensory Sural Ankle Ampltiude | 8.01 (1.55) | 8.33 (1.83)

2. Primary Outcome: Measurements of Indices of Large and Small Fiber Nerve Function Including Heart Rate Variation Measures.
Description: Quantitative Autonomic Function Tests (QAFTs) were performed. Primarily, power spectral analysis of heart rate variability (HRV) and time- and frequency-domain analyses, including measures of the sympathetic and parasympathetic control of the heart beat (R-R interval), were recorded with deep breathing, Valsalva, and standing from the sitting position maneuvers. Additionally, the sample difference of the beat to beat (NN) intervals and the TSP was calculated as well as the standard deviation of all normal R-R intervals (sdNN).
Time Frame: One year
Measure: Mean (Standard Error); unit: ms
Arm/Group | Placebo | Lovaza
Number analyzed (Participants) | 19 | 19
ms
  Resting sdNN (ms) | 31.924 (15.509) | 40.748 (16.050)
  Resting rmsSD (ms) | 28.838 (15.592) | 72.075 (30.165)
  Deep Breathing sdNN (ms) | 3.840 (10.703) | 11.637 (11.426)
  Deep Breathing rmsSD (ms) | 20.823 (2.462) | 38.136 (10.539)
  Valsalva sdNN (ms) | 0.136 (0.077) | 6.333 (13.516)
  Valsalva rmsSD (ms) | 12.752 (15.511) | 26.668 (20.514)
  Standing sdNN (ms) | 5.3786 (10.361) | 8.622 (12.080)
  Standing rmsSD (ms) | 23.725 (20.551) | 38.243 (21.850)

3. Primary Outcome: Measurements of Indices of Large and Small Fiber Nerve Function Using Vibration and Thermal Thresholds.
Description: Quantitative Sensory Tests (QSTs), including, cold sensation threshold, cold pain threshold and vibration detection threshold, were used to evaluate peripheral sensory perception.
Time Frame: One year
Measure: Mean (Standard Error); unit: °C
Arm/Group | Placebo | Omega-3-ethyl Esters 4g
Number analyzed (Participants) | 19 | 19
°C
  Cold Sensation Threshold-Finger (°C) | 0.311 (0.469) | 0.221 (0.749)
  Cold Pain Threshold-Finger (°C) | -1.167 (1.525) | -1.789 (1.882)
  Cold Sesnation Threshold-Toe (°C) | -1.169 (1.183) | -3.763 (1.647)
  Cold Pain Threshold-Toe (°C) | 5.658 (1.906) | -1.405 (2.158)
  Cold Sensation Threshold-Dorsum (°C) | -2.062 (1.484) | -3.768 (1.709)
  Cold Pain Threshold-Dorsum (°C) | 0.937 (2.215) | -1.739 (2.339)

4. Primary Outcome: Percent Change in Measurements of Indices of Large and Small Fiber Nerve Function Including Vibration Thresholds
Description: Quantitative Sensory Tests (QSTs), including vibration detection threshold, were used to evaluate peripheral sensory perception. Mean represents percent change of total group. Measurements taken at baseline and at one year.
Time Frame: One year
Measure: Mean (Standard Error); unit: % Change
Arm/Group | Placebo | Omega-3-ethyl Esters 4g
Number analyzed (Participants) | 19 | 19
% Change
  Vibration Detection Threshold-Finger (% Change) | -0.375 (0.241) | -1.102 (0.309)
  Vibration Detection Threshold-Toe (% Change) | -3.750 (5.321) | -8.169 (3.263)

5. Primary Outcome: Measurements of Indices of Large and Small Fiber Nerve Function Including Markers of Inflammation and Oxidative Stress.
Description: Oxidative stress/inflammatory markers (IL1β, IKKβ, TLR4, TNF-α, JNK1, toll-like receptor 2) were assessed through a meal challenge.
Time Frame: One year
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo | Omega-3-ethyl Esters 4g
Number analyzed (Participants) | 19 | 19
pg/ml
  IL1β (pg/ml) | 1.13 (0.21) | 1.14 (0.31)
  IKKβ (pg/ml) | 0.98 (0.16) | 0.96 (0.17)
  TLR4 (pg/ml) | 1.11 (0.18) | 1.17 (0.29)
  TNFα (pg/ml) | 1.18 (0.19) | 0.76 (0.11)
  JNK1 (pg/ml) | 0.94 (0.15) | 0.75 (0.21)
  toll-like receptor 2 (pg/ml) | 0.90 (0.12) | 0.87 (0.16)

6. Primary Outcome: Efficacy Measures Are Nerve Conduction Studies; Specifically, Increases in Conduction Velocity.
Time Frame: One Year
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Placebo | Omega-3-ethyl Esters 4g
Number analyzed (Participants) | 19 | 19
m/s
  Tibial Nerve Popliteal Conduction Velocity | 41.08 (6.58) | 37.53 (1.51)
  Median Nerve Elbow Conduction Velocity | 45.89 (1.76) | 46.74 (1.23)
  Peroneal Motor Nerve Bel. Fib. Conduction Velocity | 40.36 (1.35) | 39.96 (1.31)
  Peroneal Motor Nerve Abo. Fib. Conduction Velocity | 44.44 (3.65) | 45.00 (2.89)
  Sensory Median Nerve Wrist Conduction Velocity | 43.76 (3.08) | 46.59 (1.87)
  Sensory Ulnar Wrist Conduction Velocity | 46.94 (1.73) | 45.22 (1.75)
  Sensory Sural Ankle Conduction Velocity | 39.03 (1.61) | 38.60 (1.57)

7. Primary Outcome: Efficacy Measures Are Nerve Conduction Studies, Specifically Changes in Latency.
Time Frame: One Year
Measure: Mean (Standard Error); unit: ms
Arm/Group | Placebo | Omega-3-ethyl Esters 4g
Number analyzed (Participants) | 19 | 19
ms
  Tibial Nerve Ankle Latency | 5.08 (0.28) | 5.29 (0.31)
  Tibial Nerve Popliteal Latency | 14.65 (0.51) | 16.41 (0.66)
  Median Nerve Wrist Latency | 4.81 (1.15) | 4.56 (0.19)
  Median Nerve Elbow Latency | 9.16 (0.43) | 8.79 (0.35)
  Peroneal Motor Nerve Ankle Latency | 5.77 (0.49) | 5.24 (0.21)
  Peroneal Motor Nerve Below Fibular Latency | 13.58 (0.77) | 13.20 (0.40)
  Peroneal Motor Nerve Above Fibular Latency | 15.37 (0.95) | 14.92 (0.45)
  Sensory Median Nerve Wrist Latency | 3.48 (0.33) | 3.01 (0.16)
  Sensory Ulnar Wrist Latency | 2.51 (0.13) | 2.62 (0.11)
  Sensory Sural Ankle Latency | 3.68 (0.15) | 3.70 (0.14)

8. Primary Outcome: Efficacy Measures Are Nerve Conduction Studies, Specifically Changes in F-wave Conduction
Time Frame: One Year
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Placebo | Omega-3-ethyl Esters 4g
Number analyzed (Participants) | 19 | 19
m/s
  Tibial Nerve F-Wave Conduction | 51.14 (3.02) | 55.89 (2.45)
  Median Nerve F-Wave Conduction | 29.46 (1.09) | 29.44 (0.90)
  Peroneal Motor Nerve F-Wave Conduction | 41.96 (3.09) | 47.47 (2.49)

9. Primary Outcome: Efficacy Measures Examining Increased Vascular Response to Ischemic Block and to Local Warming at the Dorsum of the Foot.
Time Frame: One Year
Population: Measures of vascular response to ischemic block and local warming at the dorsum of the foot were not reliably collected for this assessment due to the difficulty of analysis and the inability to properly distinguish a vascular response in patients.
Arm/Group | Placebo | Omega-3-ethyl Esters 4g
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse event data was collected per individual from time of consent to 6 months after consent.
Arm/Group | Placebo | Lovaza
Serious Adverse Events (participants affected / at risk) | 4/19 | 2/19
Other Adverse Events (participants affected / at risk) | 7/19 | 8/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Lovaza (N=19)
Atypical Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Normal EKG, no evidence of myocardial infarction, normal stress test and echocardiogram and troponin normal
Head trauma due to accidental fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Patient fell and suffered bruises and cuts to her face; received more than 25 stitches and wound care to her face. Later, patient experienced vomiting and headaches and later received a CAT scan which displayed an internal head bleed due to trauma.
Hospitilization due to low blood pressure and fainting (Cardiac disorders) | 1 (1) | 0 (0) — Patient passed out in home, ER recorded BP as 63/48. During ER stay, patient had an EKG, MRI, ultrasound, and carotid doppler tests which all proved to be normal. Cause of fainting undetermined.
Overnight stay in ER for observation after experiencing chest pain (Cardiac disorders) | 1 (1) | 0 (0) — Patient seen in ER after reporting feeling pain in chest that "radiated down her arm" and some pain in her back and abdomen. A nuclear stress test was performed and patient states that no blockages were found.
Planned surgery to treat Achalasia/Esophageal motility disorder (Surgical and medical procedures) | 1 (1) | 0 (0) — Patient underwent a planned surgical procedure to treat Achalasia/Esophageal motility disorder. Procedure lasted 6 hours, and patient was under anesthesia for 7 hours. This was an in-patient procedure.
Emergency Surgery to relieve bile duct obstruction (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient went to ER reporting abdominal pain, losing 6 pounds, dark urine and clay-colored stool.CT scan found 2 stones in gallbladder - 1 occluding the common bile duct. An Endoscopic Retrograde Cholangiopancreatography removed both offending stones.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Lovaza (N=19)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient administered 5-day Z-pack; all symptoms subsided
Severe-Moderate Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2) — Patient experienced severe to moderate diarrhea which was explained as "uncontrollable" at times
Dehyrdation/Severe Vomiting/Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2) — Patient went to ER for severe dehydration (administered 2 IV bags) and nausea (given Zofran). Patient went back to ER two weeks later for similar symptoms. Dehydration most likely due to vomiting and severe diarrhea
Personal Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Patient slipped in shower and struck right elbow against the shower wall. Patient seen at ER, where x-rays revealed no abnormalities.
Dizziness/Fainting (Nervous system disorders) | 0 (0) | 1 (2) — While stopped at red light, patient reports feeling dizzy and then fainting causing her to strike another car. Bloodwork/CT done at ER with normal results. Cause of fainting undetermined.
Fainting/Dizziness (Nervous system disorders) | 0 (0) | 1 (2) — While exiting a vehicle, patient reports fainting (no dizziness reported). Cause of fainting unknown.
Eye Discharge (Eye disorders) | 0 (0) | 1 (1) — Patient reports experiencing significant increases in eye discharge. Patient reports seeing an ophthalmologist with no significant abnormalities noted.
Cranial/Facial Lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Patients reports sores on scalp and unhealing dark spots on facial skin. Patients also reports "stabbing" pain in left knee and left side of foot.
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient reports experiencing lower left quadrant pain with increased night sweats and low-grade fever. Patient seen at ER, where CAT scan revealed swollen lymph nodes in the small mesenteric bowel.
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0) — Patient reports a bacterial infection and rash on abdomen and chest. Seen at dermatologist and prescribed prescription body wash, Z-pack, and skin culture.
Personal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Rising from a seated position, patient fell. No dizziness, shortness of breath, or blurred vision noted. Patient did not receive any further medical attention.
Bladder Suspension with Sling (Surgical and medical procedures) | 1 (1) | 0 (0) — Patient underwent cystoscopy with transobturator sling. Not considered an emergency surgery.
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient suffered asthma-related bronchitis; prescribed prednisone, antibiotic, and inhaler.
Upper limb weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient reports increased arm pain/weakness bilaterally. Ordered nerve conduction study on median, ulnar, and radial nerves bilaterally resulting in otherwise normal results.
Dry/Achy Eyes (Eye disorders) | 1 (1) | 0 (0) — Patient reports experiencing increased eye strain and very dry eyes. Patient seen at ophthalmologist; prescribed artificial tears to be take Q 4 hours.
Bells Palsy (Nervous system disorders) | 1 (1) | 0 (0) — During routine physical, patient showed signs and symptoms of having Bells Palsy. Patient also reports being recently diagnosed with genital herpes. Patient prescribed metrozol pack and valtrex.
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient reports experiencing increased lower back pain. Went to ER, where x-rays revealed no significant findings. Pain attributed to soft tissue injury due to overactivity or arthritis. Received two shots of Dilaudid.
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) — Patients reports consistent higher than normal blood glucose levels. Patient instructed to continue to monitor levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No